CLINICAL TRIAL: NCT06778681
Title: Is Cortical Motor Neuron Dysfunction the Underlying Mechanism of Fatigue in Fibromyalgia?
Brief Title: Mechanism of Fatigue in Fibromyalgia and Cortical Motor Neuron Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fuat Orhun Alayoglu, Resident Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/438
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
Keywords: Fatigue; Fibromyalgia; Cortical motor neuron dysfunction; V-Wave
MeSH Terms: conditions — Fibromyalgia; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia (Experimental): Subjects with diagnosed fibromyalgia will be in this arm. Subjects will have their grip strength and 4-meter walking speed measured and will be asked to fill the fatigue severity scale.
  Subjects will be tested for v-wave during voluntary foot plantarflexion.
  Interventions: Other: Cheer
- Healthy (Experimental): Healthy subjects will be in this arm. Subjects will have their grip strength and 4-meter walking speed measured and will be asked to score the fatigue severity scale.
  Subjects will be tested for v-wave during voluntary foot plantarflexion.
  Interventions: Other: Cheer

INTERVENTIONS:
Other: Cheer — During voluntary muscle contraction subjects will be cheered with verbal encouragement ("push, push, push") and clapping.

SUMMARY:
The goal of this study is to test whether cortical motor neuron dysfunction plays a role in the pathogenesis of fatigue in fibromyalgia patients.

The main questions it aims to answer are:

Do fibromyalgia patients have lower v-wave compared to healthy subjects? Does cheering affect V-wave in fibromyalgia patients more than healthy subjects? Researchers will compare the V-waves of fibromyalgia patients with those of healthy subjects.

DETAILED DESCRIPTION:
All volunteers will first undergo the Fatigue Severity Scale (FSS) assessment, grip strength measurement, and a 4-meter walking speed test. Subsequently, V-wave recordings will be performed.

EMG and Force Data Acquisition

Surface EMG from the soleus muscle and force sensor data will be collected at a 2 kHz sampling rate using a data acquisition system (CED 3601 Power 1401 MKII digital-to-analogue converter and CED 1902 Quad System MKIII amplifier). Data analyses will be performed using Spike2 version 7.20 software.

Maximal plantar flexion will be performed against a force platform equipped with a force sensor (FC2231-0000-0100-L Compression Load Sensor, France) mounted on a wall and connected to a data acquisition device. Participants will be fixed to the examination table using a pelvic strap to prevent cranial movement during the contraction. This setup will allow real-time recording of muscle force during the 1-minute isometric contraction.

V-Wave Measurement Procedure

The procedure involves positioning participants prone on an examination table. Two self-adhesive Ag/AgCl surface electrodes (KENDALL® Coviden, Massachusetts, USA) will be placed on the belly of the left lateral soleus muscle with a 4 cm inter-electrode distance. A grounding electrode will be placed over the malleolus.

Before attaching the electrodes, any hair on the skin will be shaved, and the skin will be cleaned with alcohol wipes to remove surface oils. An ECG gel will be applied to increase skin conductivity.

For the V-wave measurement:

A cathode electrode (1 cm diameter round electrode) will be positioned over the tibial nerve in the left popliteal fossa, and an anode electrode (10x10 cm) will be placed over the suprapatellar area.

Stimulation will be delivered using a constant-current stimulator [model DS7A, Digitimer Ltd, Hertfordshire, UK] with monophasic rectangular current pulses of 1 ms duration.

The current intensity will start at 5 mA and incrementally increase. The intensity required to achieve the recruitment curve of the H-reflex and the maximum M-response (Mmax) will be determined. Supramaximal stimulation at 1.2 times the Mmax intensity will be applied to record the V-wave response.

Recording of V-Wave Responses

A one-minute fatigue protocol will be applied to see the effect of Cheer on fatigue. For this purpose, V responses will be recorded during maximum voluntary plantar flexion maintained for 60 seconds. Four V-wave responses will be recorded during the 3rd, 20th, 40th and 60th seconds of contraction. Before 60th second measurement, maximal voluntary contraction will be accompanied by verbal encouragement ("push, push, push") and clapping. Supramaximal stimulation will be given during specified times to measure v-wave.

Sample size calculation

For the V-wave measurements, repeated measures analysis of variance (ANOVA) will be used to analyze the four measurements within the two groups. Assuming a medium effect size (partial eta squared = 0.06), an alpha error level of 0.05, and a power of 0.95, the minimum required sample size was calculated to be 18 participants per group, resulting in a total of 36 participants.

The sample size calculation was performed using G*Power software version 3.1.9.4 (Franz Faul, University of Kiel, Germany).

Statistical Analysis

The normality of data distribution will be assessed using the Shapiro-Wilk test. Continuous numerical variables will be summarized as mean and standard deviation, while categorical variables will be presented as frequencies (percentages).

If the data follow a normal distribution, V-wave amplitudes will be compared using repeated measures analysis of variance (ANOVA). In cases where the analysis yields a p-value < 0.05, post-hoc pairwise comparisons will be conducted to identify differences in V-wave responses obtained during different stimulations.

If the data does not follow a normal distribution, within-group comparisons will be performed using the Friedman test and Wilcoxon test, while between-group comparisons will be performed using the Mann-Whitney U test. Post-hoc pairwise comparisons will be evaluated with Bonferroni-adjusted p-values, where a corrected p-value < 0.05 will be considered statistically significant.

All analyses will be conducted using SPSS software version 18.0.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with fibromyalgia according to acr 2016 criteria(for fibromyalgia group)
* Being healthy(for control group)
* 18-60 years old
* Volunteering
* Being female
* Right hand dominant

Exclusion Criteria:

* Presence of scars, dermatitis, or similar conditions on the skin where surface EMG electrodes will be placed.
* Diseases causing muscle and nerve dysfunction: myopathies, polyneuropathy, radiculopathy, peripheral nerve lesions such as entrapment neuropathies; central nervous system disorders such as stroke, amyotrophic lateral sclerosis, multiple sclerosis, and parkinsonism.
* Hypertension and cardiac arrhythmias.
* Other diseases with fatigue symptoms: cardiopulmonary diseases, hypothyroidism, polymyalgia rheumatica, major depression, bipolar disorder, chronic fatigue syndrome.
* Epilepsy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
V-wave | On the day of testing
  Subjects will be asked to perform voluntary foot plantar flexion. During 3rd, 20th, 40th, and 60th seconds v-wave will be measured. During the 60th second of voluntary foot plantar flexion subjects will be cheered to increase their flexion strength. V-wave/H-max ratio and V-wave amplitude changes during cheer will be compared between healthy and fibromyalgia subjects. A low ratio or amplitude will be interpreted in favor of fatigue.

SECONDARY OUTCOMES:
Fatigue severity scale | On the day of testing
  Subjects will be asked to fill in the fatigue severity scale before the study. Fatigue severity scale is scored between 1 and 7, with higher scores indicating greater fatigue.
Grip strength | On the day of testing
  Subjects will have their grip strength measured using a Jamar hand dynamometer. Results will be recorded in kilograms-force.
4m walking speed | On the day of testing
  Subjects will be asked to walk a 4-meter distance at a normal pace. They will be timed with a chronometer and walking speed will be calculated in meters/second.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)